CLINICAL TRIAL: NCT07333859
Title: Effect of Intravenous Lidocaine Infusion on Duodenal Peristalsis, Sedation Quality and Rescue Spasmolytic Requirement in ERCP Procedures: A Randomized, Double-Blind, Placebo-Controlled Study
Brief Title: Effect of IV Lidocaine on Duodenal Peristalsis and Sedation in ERCP
Acronym: LIDO ERCP
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Ankara City Hospital Bilkent (Other)
Responsible Party: Principal Investigator, Mehmet sahap, Asist Prof Dr, Ankara City Hospital Bilkent
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ERCP-LIDO-2026-01; MEHMET SAHAP (Other: ANKARA BILKENT CITY HOSPİTAL)
Record Dates: First submitted 2025-12-30; First posted 2026-01-12 (Actual); Last update posted 2026-01-12 (Actual); Status verified 2025-12

CONDITIONS: Duodenal Spasm; ERCP; Sedation
Keywords: lidocaine; Peristalsis; Intravenous Anesthesia; deep sedation; Duodenoscopy
MeSH Terms: interventions — Lidocaine; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Lidocaine Group (Experimental): 1.0 mg/kg IV bolus followed by 2.0 mg/kg/h IV infusion during the procedure.
  Interventions: Drug: Lidocaine Hydrochloride 2%; Other: 0.9 % Normal Saline
- Placebo Group (Placebo Comparator): IV bolus and infusion of 0.9% NaCl matched in volume and rate to the study drug.
  Interventions: Drug: Lidocaine Hydrochloride 2%; Other: 0.9 % Normal Saline

INTERVENTIONS:
Drug: Lidocaine Hydrochloride 2% — 1.0 mg/kg IV bolus followed by 2.0 mg/kg/h IV infusion during the procedure.
Other: 0.9 % Normal Saline — IV bolus and infusion of 0.9% NaCl matched in volume and rate to the study drug.

SUMMARY:
This study aims to evaluate the efficacy of intravenous lidocaine infusion on duodenal peristalsis during Endoscopic Retrograde Cholangiopancreatography (ERCP). The study compares lidocaine against a placebo to determine if lidocaine can reduce the need for rescue spasmolytics (hyoscine-N-butylbromide or glucagon), decrease propofol consumption, and improve hemodynamic stability.

DETAILED DESCRIPTION:
Duodenal peristalsis can hinder successful cannulation during ERCP. Traditionally, antispasmodics like hyoscine-N-butylbromide are used but have side effects. This randomized, double-blind, placebo-controlled trial includes 100 patients (ASA I-III) undergoing elective ERCP.

Patients will be randomized 1:1 into two groups:

Group L (Lidocaine): IV bolus 1.0 mg/kg before induction + 2.0 mg/kg/h continuous infusion during the procedure.

Group C (Control): Equal volume of 0.9% Saline. Primary outcome is the "Rescue Spasmolytic Requirement" based on endoscopist's evaluation. Secondary outcomes include duodenal peristalsis score (Suzuki Scale) assessed via video review by a blinded endoscopist, total propofol consumption, and recovery times.

ELIGIBILITY:
Inclusion Criteria:

* Patients scheduled for elective ERCP.

ASA Physical Status I, II, or III.

Age between 18 and 85 years.

Provided written informed consent.

Exclusion Criteria:

* Allergy to amide-type local anesthetics.

Severe hepatic or renal failure.

History of AV block or severe cardiac arrhythmia.

Pregnancy or lactation.

Chronic opioid use.

Patient refusal.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2026-02-01 (Estimated); Study Completion 2026-02-15 (Estimated)

PRIMARY OUTCOMES:
Rescue Spasmolytic Requirement Rate | Intraoperative (During the ERCP procedure, approx. 30 minutes)
  The proportion of patients requiring rescue medication (Hyoscine-N-butylbromide or Glucagon) due to severe duodenal spasm preventing cannulation.

SECONDARY OUTCOMES:
Total Propofol Consumption | Intraoperative
  Assessed using the Suzuki Scale (1=No peristalsis, 5=Severe peristalsis) via blinded video review.

IPD SHARING:
Plan to Share IPD: No
"Individual participant data will not be shared due to privacy concerns and the lack of a dedicated data management infrastructure to ensure secure anonymization.

REFERENCES:
- [Background] Suzuki M, Sekino Y, Hosono K, Kurita Y, Uechi H, Kuzuu K, Uchiyama S, Kawana K, Nagase H, Kubota K, Yoneda M, Nakajima A. Inhibitory Effect of Lidocaine on Duodenal Peristalsis During Endoscopic Retrograde Cholangiopancreatography: A Multicenter, Randomized Controlled Trial (With Video). DEN Open. 2025 Nov 27;6(1):e70252. doi: 10.1002/deo2.70252. eCollection 2026 Apr. PMID 41321955
- [Background] Abrahams M, Derby R, Horn JL. Update on Ultrasound for Truncal Blocks: A Review of the Evidence. Reg Anesth Pain Med. 2016 Mar-Apr;41(2):275-88. doi: 10.1097/AAP.0000000000000372. PMID 26866299
- [Background] Busch R, Murti K, Liu J, Patra AK, Muhammad K, Knobeloch KP, Lichtinger M, Bonifer C, Wortge S, Waisman A, Reifenberg K, Ellenrieder V, Serfling E, Avots A. NFATc1 releases BCL6-dependent repression of CCR2 agonist expression in peritoneal macrophages from Saccharomyces cerevisiae infected mice. Eur J Immunol. 2016 Mar;46(3):634-46. doi: 10.1002/eji.201545925. Epub 2016 Jan 8. PMID 26631626